CLINICAL TRIAL: NCT01225471
Title: Phase1/2 Study of Vaccination With CDCA1 Derived Epitope Peptide for HLA-A24-positive Patients With Advanced Prostate Cancer
Brief Title: Novel Peptide Vaccination for Patients With Advanced Prostate Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Iwate Medical University (Other)
Collaborators: Human Genome Center, Institute of Medical Science, University of Tokyo (Other)
Responsible Party: Departmet of Urology, Iwate Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMU-H21-40-PⅠ/Ⅱ
Record Dates: First submitted 2010-10-20; First posted 2010-10-21 (Estimated); Last update posted 2011-06-23 (Estimated); Status verified 2009-06

CONDITIONS: Prostate Cancer
Keywords: novel epitope peptide; CTL; advanced prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: CDCA1 — CDCA1-A24-56 will be administered by subcutaneously injection once every week for 3 months thereafter once two weeks. This peptide conjugated with Montanide ISA 51 as an adjuvant.

SUMMARY:
The purpose of this study is to evaluate the safety and clinical efficacy of novel peptide vaccination for advanced prostate cancer

DETAILED DESCRIPTION:
Cell division cycle associated gene 1(CDCA1) has been identified using genome-wide expression profile analysis by the use of cDNA microarray in our previous studies. We have determined the HLA-A*2402 restricted epitope peptides derived from CDCA1, CDCA1-A24-56. This epitope showed strong IFN-g production when stimulated with the appropriate targets expressed the appropriate protein and HLA-A*2402. Furthermore, when vaccinated this peptide, specific CTL was determined after the vaccination. Therefore we focused on the safety and efficacy of novel vaccination for the advanced prostate cancer patients who already showed resistance to standard hormonal therapy and chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

DISEASE CHARACTERISTICS advanced prostate cancer which already showed resistance to standard treatments

PATIENTS CHARACTERISTICS

1. Patients who showed resistance to hormonal therapy and chemotherapy
2. Histological diagnosis is adenocarcinoma
3. HLA-A*2402
4. ECOG performance status of 0 to 2
5. Age ≥ 20 years, ≤85 years
6. WBC≥ 2,000/mm³, ≤12000/mm³ hemoglobin≥ 8.0g/dl Platelet count ≥ 70000/mm³ AST, ALT ≤100 IU/l Total bilirubin ≤ 1.5 mg/dl Creatinine ≤ 1.0 mg/dl PaO2≥ 70mmHg
7. life expectancy ≥ 2months
8. Able and willing to give valid written informed consent

Exclusion Criteria:

1. Pregnancy (women of childbearing potential: Refusal or inability to use effective means of contraception)
2. Breastfeeding
3. Patients willing to childbearing ( Refusal or inability to use effective means of contraception)
4. Serious infections requiring antibiotics
5. Concomitant treatment with steroids or immunosuppressing agent
6. Other malignancy difficult to control.
7. Decision of unsuitableness by principal investigator or physician-in-charge

Ages: 20 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2009-06; Primary Completion 2011-05 (Actual); Study Completion 2012-05 (Estimated)

PRIMARY OUTCOMES:
feasibility (toxicities as assessed by NCI-CTCAE version 3) | 2 years

SECONDARY OUTCOMES:
objective response rate as assessed by RECIST criteria | 2 years
measurement of PSA | 2 years
CTL response | 2 years
CD 8 population | 2 years
change in level of regulatory T cells | 2 years
PFS and OS | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Tomoaki Fujioka, MD, PhD, Study Chair — Department of Urology, Iwate Medical University
Locations (1):
- Iwate Medical University School of Medicine, Morioka, Iwate, Japan

REFERENCES:
- [Derived] Obara W, Sato F, Takeda K, Kato R, Kato Y, Kanehira M, Takata R, Mimata H, Sugai T, Nakamura Y, Fujioka T. Phase I clinical trial of cell division associated 1 (CDCA1) peptide vaccination for castration resistant prostate cancer. Cancer Sci. 2017 Jul;108(7):1452-1457. doi: 10.1111/cas.13278. Epub 2017 Jun 23. PMID 28498618